CLINICAL TRIAL: NCT05554263
Title: Comparison of Automated Control Anesthesia and Manual Control Anesthesia Methods İn Minimal Flow Anesthesia in the Mindray A9®
Brief Title: Comparison of Automated Control Anesthesia and Manual Control Anesthesia in Minimal Flow Anesthesia
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Rezan Şerefoğlu, Research assistant, Sakarya University
Other Study IDs: Autocontrolled Anesthesia
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia; Sevoflurane; Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the introduction of technology into our lives, we come across two different anesthesia management modules in anesthesia machines. The first of these is the traditional method, the manual controlled anesthesia technique; the other is the automatic controlled anesthesia technique. In our daily practice, both anesthesia techniques can be used in patients who have undergone general anesthesia. These two techniques can be used in both high-flow anesthesia and low-flow anesthesia applications.

DETAILED DESCRIPTION:
In the manual technique, the inspired and exhaled gas concentrations are regulated by the anesthetists manually by the fresh gas flow during general anaesthesia. When administered manually, low-flow anesthesia requires the attention and time of the anesthesiologist, especially the difference between the gas concentrations set in the anesthesia machine and the respiratory system, and the delay between changes in fresh gas concentrations and the end tidal fraction (EtAA) of the anesthetic agent. The most important risks of manually controlled low-flow anesthesia are hypoxia and awareness that may occur due to low doses of inhaler anesthetic agents.

In the automatic controlled anesthesia technique, it is a method in which the values desired by the anesthetists during general anesthesia are determined at the beginning of anesthesia and automatically adjusted by the anesthesia device without any additional intervention. After intubation, anesthetists set 3 parameters on the anesthesia device: inspiratory or expiratory oxygen fraction (FiO2- End tidal O2 concentration), anesthetic agent concentration (MAC or End-tidal Anesthetic agent concentration) and fresh gas flow amount. With this method, it is aimed to provide safer and more stable anesthesia. In addition, it has been stated in many previous studies that automatic control anesthesia technique reduces anesthetic gas consumption and less anesthesiologist intervention is needed to reach target values.

In our study, we aimed to compare the safety, efficiency and cost aspects of automatic controlled anesthesia and manual control methods in achieving intraoperative target anesthetic and oxygen concentrations. We hypothesized that anesthesia applied with the end-tidal control method would have a lower cost, less workload, and similar anesthetic depth with the manual control method.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-75 year-old
* ASA 1-3
* Will undergo gynecological operation
* Expected surgery time (>1 hour)

Exclusion Criteria:

* ❖ BMI >30

  * Chronic opioid use
  * Contraindication to any of the anesthetic agents to be used
  * Neurological disorders
  * Surgery lasting <1 hour

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients scheduled for elective gynecological oncology operation under general anesthesia will be included in the study.
Study Population: Patients scheduled for elective gynecological operation under general anesthesia will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
ET-AA | 10 minutes
  searching the time needed to reach the target end tidal anesthetic agent (ET-AA) concentration and the amount of anesthetic agent consumption

SECONDARY OUTCOMES:
target values | 4 hours
  number of adjustments required to stay within target values and hemodynamic stability

CONTACTS AND LOCATIONS:
Overall Officials: Rezan Şerefoğlu, Principal Investigator — Sakarya University Research And Training hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Sakarya University Medicine Faculty Department of Anaesthesiaology and Reanimation, Sakarya
  - Sakarya University Research and Training hospital, Sakarya

REFERENCES:
- [Result] Tay S, Weinberg L, Peyton P, Story D, Briedis J. Financial and environmental costs of manual versus automated control of end-tidal gas concentrations. Anaesth Intensive Care. 2013 Jan;41(1):95-101. doi: 10.1177/0310057X1304100116. PMID 23362897
- [Result] Singaravelu S, Barclay P. Automated control of end-tidal inhalation anaesthetic concentration using the GE Aisys Carestation. Br J Anaesth. 2013 Apr;110(4):561-6. doi: 10.1093/bja/aes464. Epub 2013 Jan 4. PMID 23293274